CLINICAL TRIAL: NCT01988454
Title: Characterization of Dyslipidemia in Adolescent Obesity
Status: Completed | Type: Observational
Sponsor: Health Diagnostic Laboratory, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: R2011-2103
Record Dates: First submitted 2013-11-07; First posted 2013-11-20 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole Blood and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of this pilot study is to characterize the profile of lipoprotein, inflammatory, and metabolic markers of cardiovascular disease in obese adolescents as compared to normal-weight age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-19
* BMI ≥25 (obese) or <25 (normal weight)

Exclusion Criteria:

* Prior diagnosis of any eating disorder (e.g. anorexia or bulimia)
* Prior diagnosis of any congenital lipid disorder (e.g. familial hypercholesterolemia)
* Current use (or within past 6 months) of any lipid altering medications

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Enrollment will be representative of the ethnic population of Charlotte, NC, estimated as 50% Caucasian, 35% African American, 10% Hispanic, and 5 % other.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Comparison of biomarker profiles | Baseline
  To characterize and compare lipoprotein, inflammation and metabolic markers in obese and normal weight adolescents.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Acampora, MD, Principal Investigator
Locations (1):
- The Center for Nutrition and Preventive Medicine, Charlotte, North Carolina, United States

REFERENCES:
- [Background] Ogden CL, Carroll MD, Curtin LR, Lamb MM, Flegal KM. Prevalence of high body mass index in US children and adolescents, 2007-2008. JAMA. 2010 Jan 20;303(3):242-9. doi: 10.1001/jama.2009.2012. Epub 2010 Jan 13. PMID 20071470
- [Background] Berenson GS, Srinivasan SR, Bao W, Newman WP 3rd, Tracy RE, Wattigney WA. Association between multiple cardiovascular risk factors and atherosclerosis in children and young adults. The Bogalusa Heart Study. N Engl J Med. 1998 Jun 4;338(23):1650-6. doi: 10.1056/NEJM199806043382302. PMID 9614255
- [Background] Must A, Jacques PF, Dallal GE, Bajema CJ, Dietz WH. Long-term morbidity and mortality of overweight adolescents. A follow-up of the Harvard Growth Study of 1922 to 1935. N Engl J Med. 1992 Nov 5;327(19):1350-5. doi: 10.1056/NEJM199211053271904. PMID 1406836
- [Background] Raitakari OT, Juonala M, Viikari JS. Obesity in childhood and vascular changes in adulthood: insights into the Cardiovascular Risk in Young Finns Study. Int J Obes (Lond). 2005 Sep;29 Suppl 2:S101-4. doi: 10.1038/sj.ijo.0803085. PMID 16385760
- [Background] Superko HR. Advanced lipoprotein testing and subfractionation are clinically useful. Circulation. 2009 May 5;119(17):2383-95. doi: 10.1161/CIRCULATIONAHA.108.809582. No abstract available. PMID 19414656
- [Background] Haney EM, Huffman LH, Bougatsos C, Freeman M, Steiner RD, Nelson HD. Screening and treatment for lipid disorders in children and adolescents: systematic evidence review for the US Preventive Services Task Force. Pediatrics. 2007 Jul;120(1):e189-214. doi: 10.1542/peds.2006-1801. PMID 17606543
- [Background] Kang HS, Gutin B, Barbeau P, Litaker MS, Allison J, Le NA. Low-density lipoprotein particle size, central obesity, cardiovascular fitness, and insulin resistance syndrome markers in obese youths. Int J Obes Relat Metab Disord. 2002 Aug;26(8):1030-5. doi: 10.1038/sj.ijo.0802045. PMID 12119567
- [Background] Miyashita M, Okada T, Kuromori Y, Harada K. LDL particle size, fat distribution and insulin resistance in obese children. Eur J Clin Nutr. 2006 Mar;60(3):416-20. doi: 10.1038/sj.ejcn.1602333. PMID 16278685
- [Background] Kelishadi R, Cook SR, Amra B, Adibi A. Factors associated with insulin resistance and non-alcoholic fatty liver disease among youths. Atherosclerosis. 2009 Jun;204(2):538-43. doi: 10.1016/j.atherosclerosis.2008.09.034. Epub 2008 Oct 9. PMID 19013572